CLINICAL TRIAL: NCT03621618
Title: Clinical Assessment of Arterial Dynamic Elastance in ICU Patients, Dependent on Inotropic or Vasopressor Drugs.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 + not enough resources available
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: Eadyn project 2
Record Dates: First submitted 2018-06-28; First posted 2018-08-08 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-10

CONDITIONS: Sepsis; Cardiac Failure Acute
Keywords: vasoactive medication; dynamic arterial elastance
MeSH Terms: conditions — Sepsis | interventions — Echocardiography, Stress

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dobutamine (Other): Cardiac failure
  Interventions: Diagnostic Test: dobutamine
- norepinephrine (Other): Sepsis
  Interventions: Diagnostic Test: norepinephrine

INTERVENTIONS:
Diagnostic Test: dobutamine — evaluation of effects of dobutamine on dynamic arterial elastance in cardiac failure
  Arms: dobutamine
Diagnostic Test: norepinephrine — evaluation of effects of norepinephrine on dynamic arterial elastance in sepsis
  Arms: norepinephrine

SUMMARY:
The primary goal of the study is to determine Eadyn ( = PPV/SVV) as a functional measure of arterial load, in conjunction with other actual afterload indices, systemic vascular resistance and arterial elastance. A secondary aim is the assessment of the influences of vasopressors and inotropic drugs on Eadyn, as a parameter of ventriculo-arterial coupling.

DETAILED DESCRIPTION:
Assessment of the cardiovascular status and haemodynamics comprise directly or indirectly cardiac output, which is determined by left ventricular preload, contractility, afterload and heart rate. Various haemodynamic monitors have been introduced in anaesthesia and ICU practice, providing cardiac output either non-invasively or invasively. The combined use of arterial pressure monitoring with these devices provides insight not only in cardiac output but offers bedside assessment of most determinants of cardiovascular function. Both pulse pressure variation (PPV) and stroke volume variation (SVV) have been described as dynamic descriptors of fluid responsiveness, a measure allowing optimization of preloading conditions if haemodynamics show signals of insufficient perfusion.

Arterial load can be assessed based on a two-element Windkessel model with a static and dynamic component. The static part consists of a resistive element (systemic vascular resistance: SVR = (MAP/C0)*80, with MAP, mean arterial pressure; CO, cardiac output) and a pulsatile component (net arterial compliance C = SV/arterial pulse pressure with SV, stroke volume). Arterial elastance is considered being an integrative variable, associating both steady elements and heart rate (Ea = .9*SAP/SV with EA, arterial elastance; SAP, systolic arterial pressure). The dynamic component Eadyn is the ratio of PPV and SVV during a mechanical ventilator cycle, providing a functional assessment of ventriculo-arterial coupling.

Combined use of arterial pressure tracing (or its non-invasive surrogate) and (non-) invasive stroke volume actually may provide an interesting framework for haemodynamic monitoring and subsequent optimization in many surgical, postoperative or ICU patients. This study aims to copy as good as possible the handling and the way of management as in a clinical setting.

ELIGIBILITY:
Inclusion Criteria:

- ICU patients, treated/supported with noradrenalin or dobutamine.

Exclusion Criteria:

* Septic shock
* Aortic valve regurgitation and defect of septum
* Severe aortic sclerosis, aortic prosthesis
* Severe hypertension (MAP > 130 mmHg)
* Cardiac arrhythmia
* Tachycardia with a heart rate higher than 150 bpm
* Age below 18 or above 75 y
* Patient height below 120 cm (48") or above 230 cm (90")
* Patient weight less than 30 kg (67 lbs.) or greater than 155 kg (341 lbs.)
* Intra-aortic balloon pump

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03-31 (Actual); Primary Completion 2023-06-02 (Actual); Study Completion 2023-06-02 (Actual)

PRIMARY OUTCOMES:
Change of Dynamic Arterial Elastance (Eadyn) | baseline and from 30-90 minutes after increase with 20% of vasoactive medication and haemodynamic stabilisation
  display on the hemodynamic monitor

SECONDARY OUTCOMES:
Eadyn estimation on haemodynamic monitor | from 30 to 90 minutes after increase with 20% of vasoactive medication
  display on the hemodynamic monitor

CONTACTS AND LOCATIONS:
Overall Officials: Jan Poelaert, PhD, MD, Principal Investigator — Universitair Ziekenhuis Brussel; Michel Vervoort, IR, Study Chair — Universitair Ziekenhuis Brussel
Locations (1):
- universitair Ziekenhuis Brussel, Jette, Vlaams Brabant, Belgium